CLINICAL TRIAL: NCT00038142
Title: Randomized Phase II Study of Vincristine, Doxorubicin, Cyclophosphamide and Dexrazoxane (VACdxr) With or Without ImmTher for Newly Diagnosed High Risk Ewing's Sarcoma
Brief Title: Vincristine, Doxorubicin, Cyclophosphamide and Dexrazoxane (VACdxr) in High Risk Ewing's Sarcoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID97-198; NCI-2012-01285 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Ewing's Sarcoma
Keywords: Ewing's Sarcoma; Vincristine; Doxorubicin; Adriamycin; Rubex; Cyclophosphamide; Dexrazoxane; Zinecard; VACdxr; ImmTher
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Vincristine; Doxorubicin; Cyclophosphamide; Dexrazoxane; disaccharide tripeptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: VACdxr With ImmTher (Experimental): Chemotherapy repeated every 3 weeks for 6 cycles: Vincristine 2.0 mg/m^2 (max 2.0 mg) intravenous (IV), Doxorubicin 90 mg/m^2 IV over 30 minutes, Cyclophosphamide 2.0 g/m^2 IV daily for 2 days. Dexrazoxane 900 mg/m^2 IV (30 minutes prior to doxorubicin). ImmTher 900 mcg/m^2 IV over 1 hour every week x 50-52 weeks.
  Interventions: Drug: Vincristine; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Dexrazoxane; Biological: ImmTher
- Arm B: VACdxr (Active Comparator): Chemotherapy repeated every 3 weeks for 6 cycles: Vincristine 2.0 mg/m^2 (max 2.0 mg) IV. Doxorubicin 90 mg/m^2 IV over 30 minutes, Cyclophosphamide 2.0 g/m^2 IV daily for 2 days, Dexrazoxane 900 mg/m^2 IV (30 minutes prior to doxorubicin).
  Interventions: Drug: Vincristine; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Dexrazoxane

INTERVENTIONS:
Drug: Vincristine — 2.0 mg/m^2 (max 2.0 mg) IV x 1 repeated every 3 weeks X 6.
Drug: Doxorubicin — 90 mg/m^2 IV over 30 min x 1 repeated every 3 weeks X 6.
  Other Names: Adriamycin; Rubex
Drug: Cyclophosphamide — 2.0 g/m^2 IV daily x 2 days repeated every 3 weeks X 6.
  Other Names: Cytoxan; Neosar
Drug: Dexrazoxane — 900 mg/m^2 IV (30 min prior to doxorubicin) repeated every 3 weeks X 6.
  Other Names: DXR; Zinecard
Biological: ImmTher — 900 mcg/m^2 IV over 1 hour every week x 50-52 weeks.
  Arms: Arm A: VACdxr With ImmTher

SUMMARY:
Objectives:

1. To determine if dose intensive Vincristine, Doxorubicin, Cyclophosphamide and Dexrazoxane (VACdxr) with or without ImmTherTM can improve the 2-year disease-free survival seen with standard VAC therapy.
2. To evaluate the feasibility and describe the toxicity associated with VACdxr.
3. To evaluate the feasibility and describe the toxicity of administering ImmTherTM on a weekly basis for 50- 52 weeks.
4. To determine which therapy (VACdxr+ or VACdxr-) is worthy of further evaluation.

DETAILED DESCRIPTION:
Patients will be assigned at random (as by the toss of a coin) to receive 1 of 2 treatments.

Arm A: VACdxr will be given over 2 days through a needle in a vein. On day 1, vincristine will be given over 15 minutes, and doxorubicin will be given over 30 minutes.

Dexrazoxane will be given 30 minutes before doxorubicin; this drug protects the heart from damage by doxorubicin. Cyclophosphamide will be given once a day on days 1 and 2. This will make up 1 cycle of VACdxr treatment; the cycle will be repeated every 3 weeks for up to 6 cycles.

To prevent some side effects of VACdxr, the drugs Mesna and Neupogen/or Neulasta will also be given. Mesna helps prevent bladder damage. Neupogen is a growth factor that stimulates the body to make more white blood cells. Neulasta is a growth factor related to Neupogen.

After cycle 3, surgery may be done to remove any tumor that remains. The principal investigator will also decide whether radiation treatment should be done. If so, patients will receive radiation therapy.

Starting 1 month after all treatment is done, patients will receive ImmTher. ImmTher stimulates the body's white blood cells to attack and kill tumor cells. The drug will be given through a needle in a vein over 1 hour, every week for 1 year.

Arm B: Patients will be treated the same as patients in Arm A, except that they will not receive ImmTher.

Patients may have to stay in the hospital during VACdxr treatment and after surgery. Patients will receive ImmTher in the outpatient clinic.

Before treatment starts, patients will have a complete exam including blood and urine tests and an EKG and ECHO or multiple gated acquisition scan (MUGA) (heart function tests). X-rays and CT, MRI, bone marrow aspiration, and bone scans will be done. Women will have a pregnancy test.

After each treatment with drugs, after surgery, and after radiation treatment, patients will have checkups. These will include blood and urine tests and sometimes x-rays.

After cycle 3 of VACdxr, patients will have chest x-ray and x-ray of primary tumor. CT chest, MRI, bone marrow aspiration and bone scans will be done after 3 cycles as indicated. These tests will be done to record and measure tumors.

After treatment stops, patients will return for checkups every 3 months for 2 years.

This is an investigational study. ImmTher is an investigational agent. All other study drugs are approved by the U.S. Food and Drug Administration. As many as 104 patients will take part in the study; about 95 of these will be treated at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* High risk Ewing's Family of tumors (metastatic disease at diagnosis, humerus, femur or trunk primary, bulky primary (greater than 8 cm)), or LDH greater or equal to 900 IU/ml prior to biopsy.
* No prior chemotherapy.
* Written informed consent
* Normal cardiac function (ejection fraction greater or equal to 50%).
* Males and non pregnant females.
* Biologic age 3-60 years old.
* Adequate bone marrow function (defined as an absolute peripheral granulocyte count of>500/mm3, platelet count of >75,000/mm3, and hemoglobin >8g/dl with transfusion if required).
* Adequate renal function defined as blood urea nitrogen (BUN) <30mg% and serum creatinine <1.5 x normal for age or creatinine clearance >70.
* Patients of child bearing potential must agree to use an effective method of contraception.
* Normal hepatic function (bilirubin <1.5mg/dl, serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) <3x normal).

Exclusion Criteria: N/A

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 1997-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenie S. Kleinerman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 13, 1997 to December 7, 2009. Recruitment was done within medical clinic settings.
Pre-assignment Details: Study closed early with low recruitment due to the sponsor going out of business therefore drug no longer manufactured.
Groups:
- Arm A: VACdxr With ImmTher: Chemotherapy repeated every 3 weeks for 6 cycles: Vincristine 2.0 mg/m^2 (max 2.0 mg) intravenous (IV), Doxorubicin 90 mg/m^2 IV over 30 minutes, Cyclophosphamide 2.0 g/m^2 IV daily for 2 days. Dexrazoxane 900 mg/m^2 IV (30 minutes prior to doxorubicin). ImmTher 900 mcg/m^2 IV over 1 hour every week for 50-52 weeks.
Period: Overall Study
Arm/Group | Arm A: VACdxr With ImmTher | Arm B: VACdxr
Started | 32 | 14
Completed | 10 | 7
Not Completed | 22 | 7
Not completed — Ineligible | 1 | 0
Not completed — Progressive Disease | 11 | 7
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Unknown Reason | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: VACdxr With ImmTher | Arm B: VACdxr | Total
Number analyzed (Participants) | 32 | 14 | 46
Age, Continuous [Median (Full Range); unit: years] | 15 [4 to 50] | 17 [6 to 37] | 16 [4 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 19 | 8 | 27
Region of Enrollment [Number; unit: participants]
  United States | 32 | 14 | 46

OUTCOME MEASURES:

1. Primary Outcome: 2-year Disease-free Survival (DFS): Effect of Treatment With Combination Drugs in VACdxr Given in High Doses With or Without ImmTher to Help Participants With Ewing's Sarcoma Live Longer
Description: DFS defined as survival of participants to two years post study entry without relapse.
Time Frame: 2 years
Population: Data was not collected due to early termination of the protocol
Arm/Group | Arm A: VACdxr With ImmTher | Arm B: VACdxr
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data collected for up to 6 three-week cycles of chemotherapy then up to 30 days post drug treatment which may be received for one year if receiving ImmTher.
Description: One participant from Arm A not treated was excluded from AE reporting. Since the study regimen utilizes high dose chemotherapy, grade 4 myelosuppression (neutropenia, leukopenia, granulocytopenia, anemia and thrombocytopenia) & nausea/vomiting are expected. Constitutional symptoms (fever, chills, fatigue, headache, myalgia) are expected side effects of ImmTher, a biologic agent. A grade 4 toxicity of any of those listed expected events or hospitalizations not be reported as Serious AEs.
Arm/Group | Arm A: VACdxr With ImmTher | Arm B: VACdxr
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/14
Other Adverse Events (participants affected / at risk) | 31/31 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: VACdxr With ImmTher (N=31) | Arm B: VACdxr (N=14)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: VACdxr With ImmTher (N=31) | Arm B: VACdxr (N=14)
Abdomen Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Cramping (General disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6)
Alanine Aminotransferase/ Serum Glutamic Pyruvic Transamnase (Investigations) | 1 (1) | 0 (0)
Amylase Increase (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 23 (23) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Atrophy, Subcutaneious (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bleed Platelets Grade 3, 4 (Investigations) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Candidiasis (General disorders) | 0 (0) | 1 (1)
Cardiac Function (Cardiac disorders) | 2 (2) | 0 (0)
Cardiaovascular General (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (11) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drug Fever (General disorders) | 12 (12) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Edema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 13 (13) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fever Neutropenic (Investigations) | 17 (17) | 8 (8)
Fever Unknown Origin (General disorders) | 1 (1) | 0 (0)
Fever Without Neutropenia (General disorders) | 4 (4) | 4 (4)
Granulocytopenia (Blood and lymphatic system disorders) | 20 (20) | 10 (10)
Headache (Nervous system disorders) | 19 (19) | 3 (3)
Hematuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot Flashes (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection Neutropenia (Infections and infestations) | 4 (4) | 0 (0)
Infection Without Neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irregular Menses (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 22 (22) | 10 (10)
Lymphocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mood Alteration (Psychiatric disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis (Clinical assessment) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Nail Changes (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea Alone (Gastrointestinal disorders) | 22 (22) | 9 (9)
Neuropathy: Motor (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy: Sensor (Nervous system disorders) | 1 (1) | 1 (1)
Otitis, Middle Ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain (Nos) (General disorders) | 3 (3) | 0 (0)
Pain, Other (General disorders) | 7 (7) | 0 (0)
Pain Neuropathic (Nervous system disorders) | 1 (1) | 1 (1)
Pain, Back Other (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Platelete Increase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Rigors, Chills (General disorders) | 19 (19) | 0 (0)
Sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 14 (14) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Vascular disorders) | 23 (23) | 10 (10)
Tremors (Nervous system disorders) | 1 (1) | 0 (0)
Triglyceride, Serum Increase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal Mucositis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 21 (21) | 10 (10)
Weight Loss (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early leading to small numbers of subjects analyzed; therefore, unable to accrue required number of participants to determine statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes